CLINICAL TRIAL: NCT05535790
Title: PAX: A Randomized Single-blind Controlled Trial of the Effect of Circadian Light on Hospitalized Persons With Dementia and Older Adults With Cognitive Impairments
Brief Title: Effect of Circadian Light on Hospitalized Persons With Dementia and Older Adults With Cognitive Impairments.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: Technical University of Denmark (Other); University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SJ-899
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-08

CONDITIONS: Dementia; Cognitive Impairment
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Exposure to 24-hour LED naturalistic lighting
  Interventions: Other: Naturalistic LED light
- Control group (Sham Comparator): Exposure to standard/traditional lighting setting with fluorescent tubes
  Interventions: Other: Standard/traditional lighting

INTERVENTIONS:
Other: Naturalistic LED light — Naturalistic LED light (bright light therapy) which affects Melanopic Equivalent Daylight Illuminance.
  Arms: Intervention group
Other: Standard/traditional lighting — Standard/tradtional lighting environment with fluorescent tubes
  Arms: Control group

SUMMARY:
Light stimulates the human visual system and the biological functions in the retina, also referred to as non-visual responses, e.g. hormone production. Exposure to the correct light composition can produce acute alertness and increase good sleep quality (1).

In this study, subjects will be exposed to 24-hour LED naturalistic lighting (intervention) or traditional lighting (control) during all days of hospitalization. Subjects will be blinded to the intervention as they will not be told if they are admitted to an intervention patient room or a control patient room.

The primary outcome measure is cortisol levels measured in saliva samples. Secondary outcome measures are delirium rates, length of admission, use of constant observation, mortality and adverse advent.

It is estimated that 80 subjects will be included in the study.

DETAILED DESCRIPTION:
During hospitalization, patient rooms are often associated with poor lighting conditions, and patients are often not exposed to outdoor activities. Many patients have difficulties sleeping during hospital admission, which affects health outcomes and potentially leads to prolonged admission and rehabilitation and a higher risk of developing delirium. However, the circadian rhythm can be modified with LED light, as this technology can reach sufficient levels to affect the human melanopic equivalent daylight illuminance (Melanopic EDI). A high melanopic EDI during the day is supportive for alertness and a good night's sleep. A good night's sleep is essential to prevent the development of delirium. LED lighting, which can give melanopic EDI, is called naturalistic light (1,2).

In this study, subjects will be exposed to 24-hour LED naturalistic lighting (intervention) or traditional lighting of fluorescent tubes (control) during all days of hospitalization. Subjects will be blinded to the intervention as they will not be told if they are admitted to an intervention patient room or a control patient room. The study includes subjects who are diagnosed with dementia (mild-moderate) or older adults (+65 years) who have cognitive impairments. Subjects will be screened before inclusion using a mini-mental state examination (MMSE) (3) and clinical examination by trained specialists.

To test the effect of exposure to circadian light, the study is designed as a single-centre exploratory parallel-arm randomized controlled trial. The trial will be thoroughly reported according to the CONSORT (4) statement extended guidelines

The primary outcome measure is cortisol levels measured in saliva samples. The samples are collected two times each day during hospitalization. One sample is collected at <30 minutes after the subject has woken in the morning (during the morning cortisol peak) and one sample in the evening when the highest level is expected.

Secondary outcome measures are delirium rates, length of admission, need for escape prevention, mortality, use of antipsychotics and adverse advent e.g. patient related fall incidents. Delirium rates are collected by performing a confusion assessment method (CAM) (5) score two times a day. Additional measurements are collected in patient charts.

To reach sufficient power, we estimate that 80 subjects will be included in the study. 40 subjects are admitted to the intervention room (with naturalistic lighting), and 40 are admitted to the control room (traditional/standard lighting conditions).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a recognized dementia diagnosis by the time of admission
* Patients who, during admission, are found to have cognitive impairments
* Patients who, during admission, are found to have delirium

Exclusion Criteria:

* Patients with psychiatric conditions which in and of themselves might account for the patients' cognitive impairment will be excluded
* Inability to speak (aphasia)
* Patients with a linguistic or cultural background other than Danish
* Patients with ongoing abuse of alcohol, narcotics or sedative pharmaceutics
* Patients with impaired level of consciousness due to other causes than delirium.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Cortisol | During intervention period
  Cortisol levels measured in saliva samples

SECONDARY OUTCOMES:
Delirium | During intervention period
  Delirium measured in CAM score
Length of admission | During intervention period
  Length of admission collected from patient charts
Pharmaceutics | During intervention period
  Use of pharmaceutics during hospitalization. Collected from patient charts.
Mortality | During intervention period
  Mortality rates collected from patient charts
Adverse advent | During intervention period
  Adverse advent, e.g. patient related fall incidents, collected from patient charts
Constant observation | During intervention period
  Need of constant observation from health professionals, collected from patient charts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Figueiro MG, Nagare R, Price L. Non-visual effects of light: how to use light to promote circadian entrainment and elicit alertness. Light Res Technol. 2018;50(1):38-62. doi: 10.1177/1477153517721598. Epub 2017 Jul 25. PMID 30416392
- [Background] Figueiro MG. Light, sleep and circadian rhythms in older adults with Alzheimer's disease and related dementias. Neurodegener Dis Manag. 2017 Apr;7(2):119-145. doi: 10.2217/nmt-2016-0060. Epub 2017 May 23. PMID 28534696
- [Background] Creavin ST, Wisniewski S, Noel-Storr AH, Trevelyan CM, Hampton T, Rayment D, Thom VM, Nash KJ, Elhamoui H, Milligan R, Patel AS, Tsivos DV, Wing T, Phillips E, Kellman SM, Shackleton HL, Singleton GF, Neale BE, Watton ME, Cullum S. Mini-Mental State Examination (MMSE) for the detection of dementia in clinically unevaluated people aged 65 and over in community and primary care populations. Cochrane Database Syst Rev. 2016 Jan 13;2016(1):CD011145. doi: 10.1002/14651858.CD011145.pub2. PMID 26760674
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 Statement: updated guidelines for reporting parallel group randomised trials. BMC Med. 2010 Mar 24;8:18. doi: 10.1186/1741-7015-8-18. PMID 20334633
- [Background] Wei LA, Fearing MA, Sternberg EJ, Inouye SK. The Confusion Assessment Method: a systematic review of current usage. J Am Geriatr Soc. 2008 May;56(5):823-30. doi: 10.1111/j.1532-5415.2008.01674.x. Epub 2008 Apr 1. PMID 18384586